CLINICAL TRIAL: NCT05151601
Title: The Effect of a Combination of Human Milk Oligosaccharides (HMOs) and Probiotics on Behavioural Change in Children With Autism Spectrum Disorder (ASD).
Brief Title: Combined Human Milk Oligosaccharides (HMOs) and Probiotics Intervention for Children With Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11-30-Auts
Record Dates: First submitted 2021-10-17; First posted 2021-12-09 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-02

CONDITIONS: Autism Spectrum Disorder; Neurodevelopmental Disorders; Anxiety
Keywords: Gut microbiome; Behaviour
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders; Anxiety Disorders; Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be recruited into a two-phase project. Phase 1A: an 8-week double-blinded, placebo-controlled, randomised trial. Participants child will be randomised to one of groups 1) treatment (HMOs/Probiotic group) or 2) control group (placebo product).
  Phase 1B: is an 8-week open-label trial. All children who successfully complete phase 1A will be recruited into phase 1B. All participants in phase 1B will receive the treatment product (HMOs/probiotics).
  Follow up will occur at week 8 and week 17.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMOs + Probiotics (Experimental): Dosing: A total daily dose of 2 x sachets (6g/day)
  Product Comprised of:
  1. 2.5g of a proprietary blend of human milk oligosaccharides combined with
  2. 20 billion CFUs of a mixture of Lactobacillus rhamnosus, Lactobacillus plantarum, Bifidobacterium animalis spp. lactis, and Bifidobacterium longum.
  Mode of administration: oral.
  Interventions: Dietary Supplement: Experimental
- Placebo (Placebo Comparator): Dosing: A total daily dose of 2 x sachets (6g/day)u (8 weeks of phase 1A). Product: powdered maltodextrin. Mode of administration: oral.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Experimental — 2 x sachets per day
  Arms: HMOs + Probiotics
Other: Placebo — 2 x sachets per day
  Arms: Placebo

SUMMARY:
This research project will investigate if a supplement containing a unique combination of prebiotics and probiotics can influence behaviour in children diagnosed with autism spectrum disorder. The study will use a combination of human milk oligosaccharides (HMOs, prebiotics) and probiotics as an oral powder.This clinical trial will have two consecutive phases. Phase 1A is an 8-week randomised, double-blinded, placebo-controlled trial. Participants will be recruited and randomised (1:1) to receive either the investigational product (treatment group, n=30) or the placebo (control group, n=30). Phase 1B is an 8-week open-label study. All participants that complete Phase 1A will move into Phase 1B (n=60). This allows all participants to receive the investigational product and will provide additional information on increased duration of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 5.00 years to 12.99 years.
2. A confirmed diagnosis of ASD or Pervasive Developmental Disorders (PDD) including autistic disorder, Asperger's disorder (AS); PDD not otherwise specified (PDD-NOS); and atypical autism.

Exclusion Criteria:

1. Organic GI disorders such as inflammatory bowel disease, coeliac disease, eosinophilic disorders, or current infection of the GI tract.
2. Bowel surgery or short bowel syndrome
3. Participants who have a diagnosed cow milk protein allergy.
4. Participants who suffer from the conditions listed below or who are taking any of the following medications or supplements:

   * antibiotics or antifungals in the last two months
   * probiotic supplements in the last two months
   * immunocompromised or severely ill
   * genetic disorders (e.g. Fragile X Syndrome)
   * chronic health conditions such as diabetes, heart disease or an eating disorder.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Behaviour change | Baseline, Phase IA midpoint (week 4) and post-Phase 1A(week 8/9), post-Phase 1B (week 17/18)
  Changes in behavioural symptoms as measured by the Irritability sub-scale of the Aberrant Behavior Checklist - Community (Version 2) (I-ABC). The ABC 58-item parent-rated questionnaire and consists of five subscales, including: 1) irritability (15 items); 2) lethargy/social withdrawal (16 items); 3) stereotypic behaviour (7 items); 4) hyperactivity/noncompliance (16 items); and 5) inappropriate speech (4 items). Each item is scored as 0=never a problem, 1=slight problem, 2=moderately serious problem, or 3=severe problem. The score range is 0-174, with a higher score indicating greater severity or difficulties.
Behaviour Change | Baseline, Phase 1A midpoint (week 4) and post-Phase 1A (week 8/9)
  Changes in behavioural symptoms as measured by the Home Situations Questionnaire - Autism Spectrum Disorder (HSQ-ASD). The HSQ-ASD is a 24-item, parent-rated measure of non compliant behaviour in children with ASD. The scale yields per-item mean scores of 0 to 9, with higher scores indicating greater noncompliance.
Behaviour Change | Baseline and post-Phase 1A (week 8/9)
  Changes in parent/guardian targeted behaviours as measured by the Parent Targeted Symptom Visual Analogue Scale (PTSVAS). The PTSVAS tool requests parents/guardians report their top three (3) target behaviours (behaviours of concern) on a Visual Analogue Scale (VAS). The VAS is a horizontal line of 100mm in length, with each end defined as the extreme limits of the behaviour of concern ("best" to "worst"), to be measured from left to right. The parents will score the behaviour by placing a mark on the VAS at baseline and post-intervention. Each mark will be measured on the scale of 0-100mm and the change from baseline to post-intervention noted.

SECONDARY OUTCOMES:
Change in GI Symptom Severity | Baseline and post-Phase 1A (week 8/9)
  Change in GI symptom severity as measured by the 6-item gastrointestinal severity index (6-GSI). The 6-GSI assesses each GI symptom using a Likert scale of 0-2 (0 = nil/mild/infrequent; 1 = moderate/occasional; 2 = severe/frequent). Score range 0-12. Mild GI issues are defined as a score of under three and moderate or severe GI issues defined as a score of three or above.
Change in the Gut Microbiome | Baseline and post-Phase 1A (week 8/9)
  This is an explorative outcome to compare and characterise changes in gut (stool) micorbiome between treatment groups. Change or trends (diversity, bacterial species, metabolite potential) in the gut microbiome as analysed using stool shotgun metagenomic sequencing.
Change in Anxiety Levels | Baseline and post-Phase 1A (week 8/9)
  Change in anxiety levels as measured by the Parent Rated Anxiety Scale - Autism Spectrum Disorder (PRAS-ASD) questionnaire. This is a 25-item tool using a Likert scale of 0-3 (0=none; 1=mild; 2=moderate; 3=severe). Score range 0-75, with higher scores indicating greater levels of anxiety.
Change in Quality of Life | Baseline and post-Phase 1A (week 8/9)
  Quality of life (QoL) measured by the Quality of life Autism (QoLA) questionnaire. The QoLA is a 48-item questionnaire divided into 2 subsets (Part A and Part B). The QoLA utilises a 5-point scale (0-4). Possible scores range from 48-240, with higher scores equating to higher perceived QoL.
Change in Stool Consistency | Baseline, Phase A1 midpoint (week 4), and post-Phase 1A (week 8/9), post-Phase 1B (week 17/18) .
  Change in Stool consistency as measured by the Bristol Stool Chart (BSC, paediatric version)
Change in stool short chain fatty acids levels | Baseline and post-Phase 1A (weeks 8/9)
  Change in stool short chain fatty acids levels as measured using gas chromatography with flame ionisation detection (GC-FID)
Change in urinary serotonin concentration | Baseline and post-Phase 1A (weeks 8/9)
  Change in concentrations of the urinary serotonin metabolite, 5-Hydroxyindoleacetic acid as measured using a double solvent front extraction, followed by reversed phase High Performance Liquid Chromatography (HPLC) with electrochemical detection (ECD)
Change in salivary cortisol levels | Baseline and post-Phase 1A (weeks 8/9)
  Change to salivary cortisol levels as measured using the Elecsys® Cortisol II assay

CONTACTS AND LOCATIONS:
Overall Officials: Peter SW Davies, PhD, Principal Investigator — The University of Queensland
Locations (1):
- University of Queensland, Child Health Research Centre, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
IPD is the intellectual property of the funding industry partner.